CLINICAL TRIAL: NCT00665392
Title: Induction Chemotherapy With Cetuximab, Docetaxel, Cisplatin, and Fluorouracil (ETPF) in Patient With Resectable Stage III-IV Squamous Cell Carcinoma of the Oropharynx
Brief Title: Cetuximab and Combination Chemotherapy in Patients With Stage III-IV Resectable Oropharynx Cancer
Acronym: ECHO-07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593027; GERCOR-ECHO-07-1 (Other: GERCOR); 2007-002116-25 (EudraCT Number); EU-20838 (Registry Identifier: EU Clinical Trials Register); MERCK-GERCOR-ECHO-07-1 (Other: GERCOR)
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cisplatin; Docetaxel; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab (Experimental): Cetuximab by intravenous (IV) infusion over 1-2 h on day
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil; Drug: Cetuximab

INTERVENTIONS:
Drug: cisplatin — 75 mg/m², day 1. 3 cycles
Drug: docetaxel — 75 mg/m² Day 1. 3 cycles
Drug: fluorouracil — 750 mg/m² day 1 to day 5. 3 cycles
Drug: Cetuximab — 400 mg/m² Day 1, 250 mg/m² Day 8 and Day 15. 3 cycles.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with cetuximab may kill more tumor cells.

PURPOSE: This phase II clinical trial is studying how well cetuximab given together with combination chemotherapy works in treating patients with stage III or stage IV oropharynx cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete clinical response rate at 3 months in patients with stage III or IV nonmetastatic squamous cell carcinoma of the oropharynx treated with cetuximab, docetaxel, cisplatin, and fluorouracil.

Secondary

* To determine the rate of tumor response.
* To determine progression-free and overall survival.
* To determine the rate of complete pathological response.
* To assess the tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15; docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1; and fluorouracil IV continuously on days 1-5. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 2 months for 1 year and every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oropharynx

  * Stage III (T3 or T1-2, N1-2, M0) or nonmetastatic stage IV (T4 or T1-3, N3, M0) disease
  * Resectable disease
* Measurable or evaluable disease
* Tumor tissue available

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-1
* ANC ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 9 g/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 60 mL/min
* AST and ALT < 5 times ULN
* Bilirubin < 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Affiliated with social security (including CMU)

Exclusion criteria:

* Cardiovascular accident (myocardial infarction, cerebral vascular accident) within the past 6 months
* Serious and/or uncontrolled cardiac or respiratory disease (pulmonary fibrosis, interstitial pneumopathy)
* Other cancer within the past 5 years except for resected skin cancer, localized cutaneous or totally resected melanoma, or resected carcinoma in situ of the cervix
* Auditory condition precluding the use of cisplatin
* Contraindication due to psychological, social, or geographical reasons that may impede proper monitoring of treatment
* Persons under guardianship or trusteeship, or prisoners of law

PRIOR CONCURRENT THERAPY:

* No prior treatment, including chemotherapy or radiotherapy
* No concurrent phenytoin, live attenuated vaccines, or parenteral aminoglycosides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2013-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lacau Saint Guily, MD, Principal Investigator — Hopital Tenon
Locations (8):
- France (8):
  - Hôpital Simone Veil, Montmorency
  - Hôpital Privé St Joseph, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Tenon, Paris
  - centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre René Huguenin, Saint-Cloud
  - Hopital Foch, Suresnes

REFERENCES:
- [Result] Chibaudel B, Lacave R, Lefevre M, Soussan P, Antoine M, Perie S, Belloc JB, Banal A, Albert S, Chabolle F, Ceruse P, Baril P, Gatineau M, Housset M, Moukoko R, Benetkiewicz M, de Gramont A, Bonnetain F, Lacau St Guily J. Induction therapy with cetuximab plus docetaxel, cisplatin, and 5-fluorouracil (ETPF) in patients with resectable nonmetastatic stage III or IV squamous cell carcinoma of the oropharynx. A GERCOR phase II ECHO-07 study. Cancer Med. 2015 May;4(5):721-31. doi: 10.1002/cam4.408. Epub 2015 Feb 14. PMID 25684313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2008 to April 2013, 42 patients were enrolled. This study was conducted in France, in 9 active centers: Hospital Tenon, HEGP, Hospital Bichat, GH St Joseph Paris, Hospital Foch Suresnes, CH Lyon Sud, Hospital Delafontaine St Denis, Centre René Huguenin St Cloud et Hospital Simone Veil Montmorency.
Pre-assignment Details: The main inclusion criteria: Previously untreated, resectable stage III (T3 or T1 - 2N1 - 2M0) to IVB (T4 or T1 -3N3M0) SCCHN of the oropharynx, measurable or evaluable disease, WHO performance status ≤ 1, adequate hematologic, renal and liver functions.
  The main exclusion criteria: uncontrolled cardiac or other disease, hearing impairment
Groups:
- ETPF Adminstration: cisplatin: 75 mg/m², day 1. 3 cycles
  docetaxel: 75 mg/m² Day 1. 3 cycles
  fluorouracil: 750 mg/m² day 1 to day 5. 3 cycles
  Cetuximab: 400 mg/m² Day 1, 250 mg/m² Day 8 and Day 15. 3 cycles.
Period: Overall Study
Arm/Group | ETPF Adminstration
Started | 42
Completed | 41
Not Completed | 1
Not completed — not treated | 1

BASELINE CHARACTERISTICS:
Population: 42 patients enrolled and 41 treated. Forty-one patients (mITT population) started induction therapy. One patient did not receive an intended treatment due to investigator decision to replace cisplatin by carboplatin and not to administer cetuximab.
Arm/Group | Cetuximab
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 34
Region of Enrollment [Number; unit: participants]
  France | 42
Grade of differentiation [Number; unit: participants]
  Well | 17
  Moderate | 18
  Poor or undifferentiated | 4
  Missing | 3
Primary tumor localization [Number; unit: participants]
  Anterior | 3
  Lateral (tonsillar area) | 37
  Posterior | 1
  Superior | 1
T-stage [Number; unit: participants] — Classification for Oropharyngeal - T for Primary tumor TX Primary tumor cannot be assessed T0 No evidence of primary tumor Tis Carcinoma in situ T1 Tumor ≤2 cm in greatest dimension T2 Tumor >2 cm but not more than 4cm in greatest dimension T3 Tumor >4 cm in greatest dimension or extension to lingual surface of the epiglottis T4a Moderately advanced, local disease T4b Very advanced, local disease
  participants
    T2 | 13
    T3 | 24
    T4 | 5
N-stage [Number; unit: participants] — N for Regional lymph nodes N0 No regional lymph node metastasis N1 Metastasis in a single ipsilateral lymph node ≤3 cm in greatest dimension N2 Metastasis in a single ipsilateral lymph node >3 cm but not more than 6cm in greatest dimension; or in multiple ipsilateral lymph nodes, none >6cm in greatest dimension; or in bilateral or contralateral lymph nodes, none >6cm in greatest dimension N3 Metastasis in a lymph node >6cm in greatest dimension
  participants
    N0 | 5
    N1 | 9
    N2 | 27
    N3 | 1
Cancer Staging at the inclusion [Number; unit: participants] — Patient with resectable stade III (T3 or T1 - 2N1 - 2M0) to IVB (T4 or T1- 3N 3M0).
  Anatomic stage/prognostic groups at the inclusion. Stade III is the best pronostic than stade IV.
  participants
    III | 32
    IV | 10
Lip mobility [Number; unit: participants]
  Normal | 40
  Decreased | 2
Trismus [Number; unit: participants]
  Yes | 5
  No | 37
Creatinine clearance (mL/min) [Number; unit: participants]
  < 60 | 1
  60 -120 | 31
  > 120 | 8
  Missing | 2
Albuminemia (g/L) [Number; unit: participants]
  < 40 | 8
  ≥ 60 | 14
  Missing | 20
Life style risk factors [Number; unit: participants]
  Alcohol | 3
  Tobacco | 8
  Alcohol + Tobacco | 25
  None | 6
HPV 16 status [Number; unit: participants] — human papillomavirus type 16 status
  participants
    Positive | 17
    Negative | 25
ECOG performance status [Number; unit: participants] — The ECOG Performance Status is a method to assess the functional status of a patient.
  * ECOG PS 0 : Fully active, able to carry on all pre-disease performance without restriction
  * ECOG PS 1 : Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  participants
    ECOG - PS=0 | 33
    ECOG - PS=1 | 8
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Radiological Complete Clinical Response (crCR) Rate at 3 Months
Description: The evaluation of tumor response rate was assessed by computed tomography scan of the neck and chest at Baseline, then at 3 months from inclusion using RECIST1.0 criteria and clinical examination
Time Frame: at 3 months after ETPF combination
Measure: Number; unit: participants
Groups:
- ETPF Administration: cisplatin: 75 mg/m², day 1. 3 cycles
  docetaxel: 75 mg/m² Day 1. 3 cycles
  fluorouracil: 750 mg/m² day 1 to day 5. 3 cycles
  Cetuximab: 400 mg/m² Day 1, 250 mg/m² Day 8 and Day 15. 3 cycles.
Arm/Group | ETPF Administration
Number analyzed (Participants) | 41
participants
  Tumor response Rate - Tumor | 9
  Tumor response rate - node | 8
  Tumor response rate - Tumor and node | 4

2. Secondary Outcome: Complete Clinical Response (cCR)
Description: Clinical complete response (cCR) is defined by:
  * Disappearance of all clinical evidence of visible tumor,
  * Disappearance of all palpable residual infiltration,
  * Disappearance of all evidence of residual visible tumor on CT scan in pharynx and parapharyngeal space,
  * Complete symmetric remobilization of the tongue and amygdala.
  * Disappearance of pre-existing trismus.
  * Negative control biopsy.
  The evaluation of tumor response rate was assessed by computed tomography scan of the neck and chest at Baseline, then at 3 months from inclusion using RECIST1.0 criteria and clinical examination
Time Frame: at 3 months
Measure: Number; unit: participants
Arm/Group | ETPF Administration
Number analyzed (Participants) | 41
participants
  Tumor response rate - tumor | 17
  Tumor response rate - node | 15
  Tumor response rate - Tumor and node | 13

3. Secondary Outcome: The 2-year Estimated Overall Survival (OS) Rate
Description: 2-year OS measured survival at 2 years from randomization.
Time Frame: 2 years
Population: Median OS was not achieved. The 2-year estimated rate is given.
Measure: Number; unit: percentage of participants
Arm/Group | ETPF Administration
Number analyzed (Participants) | 41
percentage of participants | 82

4. Secondary Outcome: Pathologic Response
Description: On primary tumor resected : measure of persistence or not of tumoral lesion, histological type, size and quality of the excision piece
  A pathological complete response is defined as no viable tumour cells detected on histological examination post surgery.
Time Frame: after surgery of the primary tumor
Population: Pathological response is evaluable in patients with tumor surgical resection only
Measure: Number; unit: participants
Arm/Group | ETPF Administration
Number analyzed (Participants) | 22
participants | 9

5. Secondary Outcome: The 2-year Estimated Progression-free Survival (PFS)
Description: 2-year PFS measured survival at 2 years from randomization.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | ETPF Administration
Number analyzed (Participants) | 41
percentage of participants | 64

6. Secondary Outcome: Complete Radiological Response (rCR)
Description: Radiological response is defined according to RECIST 1.0 criteria:
  * Complete response (CR): disappearance of all target lesions
  * Partial response (PR): at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter,
  * Progressive disease (PD): at least a 20% increase in the sum of the longest diameter of target the appearance of one or more new lesions,
  * Stable disease (SD): neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started
Time Frame: At 3 months after the end of 3 cycles of the ETPF combination
Population: Patients in the mITT population who received ETPF
Measure: Number; unit: participants
Groups:
- ETPF Administration: Treatment consisted of cetuximab by intravenous (IV) infusion over 1-2 h on days 1, 8, and 15 (loading dose of 400 mg/m2 on day 1, then 250 mg/m2 weekly) followed the same day by docetaxel and cisplatin both given as a
  1h IV infusion (at a 75 mg/m2 dose) and by 5-FU IV infusion on days 1-5 (at a 750 mg/m2 dose per day). Treatment was given every 3 weeks for a maximum of three cycles.
Arm/Group | ETPF Administration
Number analyzed (Participants) | 41
participants
  Tumor response rate - Tumor | 14
  Tumor response rate - Node | 8
  Tumor response rate - Tumor and node | 4

7. Other Pre Specified Outcome: Biomarkers Analysis - HPV Genotyping
Time Frame: correlative studies investigating HPV status in tumor and blood samples obtained prior to and after induction therapy were done for exploratory purposes as planned in the protocol
Measure: Number; unit: participants
Arm/Group | ETPF Administration
Number analyzed (Participants) | 42
participants
  HPV16 - Positive | 17
  HPV16 - Negative | 25

ADVERSE EVENTS:
Time Frame: Until 1 month after the last administration
Description: Adverse events (AE) were collected during induction treatment and follow-up visit (1 month).Toxicity evaluation was carried out according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v3.0)
Arm/Group | ETPF Administration
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETPF Administration (N=41)
Hypovolaemia (Vascular disorders) | 1
Orthostatic hypotension (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3 — grade 3
Acute pancreatitis (Hepatobiliary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Febrile aplasia (Infections and infestations) | 2
sepsis (Infections and infestations) | 1
Febrile neutropenia (Infections and infestations) | 1
Infection at the portacath site (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETPF Administration (N=41)
Neutropenia (Blood and lymphatic system disorders) | 18
Anemia (Blood and lymphatic system disorders) | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Creatinine (Blood and lymphatic system disorders) | 9
Neuropathy peripheral (Nervous system disorders) | 4
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Stomatitis (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 27
Acne (Skin and subcutaneous tissue disorders) | 18
Febrile neutropenia (Infections and infestations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No